CLINICAL TRIAL: NCT03857425
Title: Helicobacter Pylori Eradication With Clostridum Butyricum Capsule and Bacillus Coagulans Tablets
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Xijing Hospital of Digestive Diseases (Other)
Responsible Party: Principal Investigator, Yongquan Shi, Principal Investigator, Clinical Professor, Xijing Hospital of Digestive Diseases
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KY20192009-F-1
Record Dates: First submitted 2019-02-26; First posted 2019-02-28 (Actual); Last update posted 2019-09-25 (Actual); Status verified 2019-02

CONDITIONS: Gastritis; H Pylori Infection; Dyspepsia
Keywords: Gastritis; H Pylori Infection
MeSH Terms: conditions — Gastritis; Dyspepsia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Clostridum Butyricum Capsule (Experimental): Clostridum Butyricum Capsule 3*420mg, twice daily for 8 weeks
  Interventions: Drug: Clostridum Butyricum Capsule
- Bacillus Coagulans Tablets (Experimental): Bacillus Coagulans Tablets 3*350mg, three times daily for 8 weeks
  Interventions: Drug: Bacillus Coagulans Tablets
- Clostridum Butyricum Capsule plus Bacillus Coagulans Tablets (Experimental): Clostridum Butyricum Capsule 3*420mg, twice daily for 8 weeks and Bacillus Coagulans Tablets 3*350mg, three times daily for 8 weeks
  Interventions: Drug: Clostridum Butyricum Capsule plus Bacillus Coagulans Tablets

INTERVENTIONS:
Drug: Clostridum Butyricum Capsule — Clostridum Butyricum Capsule 3*420mg,twice daily for 8 weeks
  Arms: Clostridum Butyricum Capsule
Drug: Bacillus Coagulans Tablets — Bacillus Coagulans Tablets 3*350mg, three times daily for 8 weeks
  Arms: Bacillus Coagulans Tablets
Drug: Clostridum Butyricum Capsule plus Bacillus Coagulans Tablets — Clostridum Butyricum Capsule 3*420mg, twice daily for 8 weeks and Bacillus Coagulans Tablets 3*350mg, three times daily for 8 weeks
  Arms: Clostridum Butyricum Capsule plus Bacillus Coagulans Tablets

SUMMARY:
This study aims at evaluating efficacy Clostridum Butyricum Capsule and Bacillus Coagulans Tablets in H. pylori eradication. It is hypothesized that Clostridum Butyricum Capsule , Bacillus Coagulans Tablets monotherapy or Clostridum Butyricum Capsule plus Bacillus Coagulans may have some positive effect on H. pylori eradication.

DETAILED DESCRIPTION:
The study will include three phases: screening, treatment and follow-up. Screening: during this phase subjects eligibility will be evaluated after informed consent signature. Endoscopy and Urea Breath test will be performed in addition to the baseline routine evaluations.

Treatment: Subjects are randomly assigned to treatment and will be treated for 8weeks.

Follow-up: includes one visits. Eradication of H. Pylori will be confirmed through urea breath test(UBT).

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18~70,both gender.
2. Patients with upper gastrointestinal symptoms and with documented H.pylori infection.
3. Patients are willing to receive eradication treatment.
4. Women are eligible if they are not pregnant or nursing, and if they are of childbearing potential they are required to use medically acceptable contraception for the duration of the study and 30 days thereafter.

Exclusion Criteria:

1. Patients are excluded if they have previously used antibiotics to eradicate adequately recorded infection with H. pylori.
2. Contraindications to study drugs.
3. Substantial organ impairment, severe or unstable cardiopulmonary or endocrine disease.
4. Constant use of anti-ulcer drugs ( including taking proton-pump. inhibitors(PPI) within 2 weeks before the [13C] urea breath test), antibiotics or bismuth complexes (more than 3 times /1 month before screening).
5. Pregnant or lactating women.
6. Patients were diagnosed with gastroduodenal ulcer and MALT lymphoma.
7. Underwent upper gastrointestinal Surgery.
8. Patients with Barrett esophageal or highly atypical hyperplasia, have symptom of dysphagia.
9. Evidence of bleeding or iron efficiency anemia.
10. A history of malignancy.
11. Drug or alcohol abuse history in the past 1 year.
12. Systemic use of corticosteroids, non steroidal anti-inflammatory drugs, anticoagulants, platelet aggregation inhibitors (except the use of aspirin for less than 100 mg/d).
13. Enrolled in other clinical trials in the past 3 months.
14. Patients who has psychological problem or poor compliance.
15. Refuse to sign informed consent.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2019-09-15 (Actual)

PRIMARY OUTCOMES:
helicobacter pylori eradication H.pylori eradication | 8 weeks
  Rate of H.pylori eradication Assessed by urea breath test，rapid urease test or helicobacter pylori stool antigen test after the end of treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Xijing Hosipital of Digestive Disease, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhang J, Guo J, Li D, Chen M, Liu J, Feng C, He Q, Zhao J, Zhang L, Chen J, Shi Y. The efficacy and safety of Clostridium butyricum and Bacillus coagulans in Helicobacter pylori eradication treatment: An open-label, single-arm pilot study. Medicine (Baltimore). 2020 Nov 6;99(45):e22976. doi: 10.1097/MD.0000000000022976. PMID 33157939